CLINICAL TRIAL: NCT00403637
Title: A Randomized, Double-blind, Double-dummy, Active (Formoterol 12 µg b.i.d) and Placebo Controlled, Multi-center, 5 Period Crossover Study to Assess the Bronchodilatory Efficacy and Safety of Single Doses of Indacaterol 150 µg, 300 µg and 600 µg Delivered Via Single Dose Dry Powder Inhaler (SDDPI) vs. Placebo in Patients With Persistent Asthma
Brief Title: Efficacy and Safety of Single Doses of Indacaterol Delivered Via a Single Dose Dry Powder Inhaler (SDDPI) Compared to Placebo in Patients With Persistent Asthma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: CQAB149A2228
Record Dates: First submitted 2006-11-06; First posted 2006-11-27 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Asthma
Keywords: Asthma, indacaterol, long acting β2-agonist
MeSH Terms: conditions — Asthma

INTERVENTIONS:
Drug: indacaterol maleate

SUMMARY:
The study is designed to obtain safety and efficacy data on three dose levels of indacaterol when delivered via an SDDPI in patients with persistent asthma. All patients will receive 1 day of treatment with each of the following: indacaterol 150 µg, indacaterol 300 µg, indacaterol 600 µg, placebo, and formoterol. Each treatment day will be followed by a washout-period of 1 week

ELIGIBILITY:
Inclusion Criteria:

* Males and females 12 - 75 years of age with a diagnosis of persistent asthma
* Daily treatment with a bronchodilator and daily dose of at least 100 µg beclomethasone dipropionate or equivalent
* FEV1 at Visit 1 at least 50% of the predicted normal value
* FEV1 reversibility at least 15%

Exclusion Criteria:

* Use of tobacco products within 6 months prior to Visit 1 or a smoking history of more than 10 pack years
* Chronic Obstructive Pulmonary Disease (COPD)
* Seasonal allergy where asthma is likely to deteriorate during the period of the study
* Emergency room treatment for an acute asthma attack within the previous 6 weeks or hospitalized within the previous 6 months
* A respiratory tract infection within the previous 6 weeks Other protocol-defined exclusion criteria may apply

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2006-11; Primary Completion 2007-02 (Actual); Study Completion 2007-02

PRIMARY OUTCOMES:
Lung function measured 24 hours after having taken medication, by a special test called "forced expiratory volume in 1 second "(FEV1)

SECONDARY OUTCOMES:
FEV1 at time points 30 min, 1, 2 and 4 h post-dose
Percent change in FEV1 at time points 30 min, 1, 2 and 4 h, 23 h 10 min and 23 h 45 min post dose
Forced vital capacity (FVC) at time points 30 min, 1, 2 and 4 h, 23 h 10 min and 23 h 45 min post dose

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Novartis
Locations (5):
- United States (5):
  - Colorado Allergy and Asthma Centres, P.C., Denver, Colorado
  - Northeast Medical Research Associates, Inc., North Dartmouth, Massachusetts
  - Clinical Research Institute, Minneapolis, Minnesota
  - The Clinical Research Center, St Louis, Missouri
  - North Carolina Clinical Research, Raleigh, North Carolina